CLINICAL TRIAL: NCT00629382
Title: Dispositivo Adsorbente Con Polymyxina B Immobilizzata Nello Shock Settico - Studio Clinico Randomizzato e Prospettico, Multicentrico
Brief Title: Early Use of Polymyxin B Hemoperfusion in Abdominal Sepsis
Acronym: EUPHAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Bortolo Hospital (Other)
Responsible Party: Claudio Ronco, MD, International Renal Research Institute Vicenza (IRRIV),
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TM05
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-04

CONDITIONS: Gram-Negative Bacterial Infections; Sepsis; Septic Shock
Keywords: abdominal sepsis; abdominal surgery; septic shock; polymyxin B; hemoperfusion; Endotoxins
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Sepsis; Shock, Septic; Intraabdominal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Polymyxin B immobilized fiber column; Other: Conventional medical therapy in the ICU
- 2 (Other)
  Interventions: Other: Conventional medical therapy in the ICU

INTERVENTIONS:
Device: Polymyxin B immobilized fiber column — Hemoperfusion with PMX will be performed in ICU. The 1st PMX treatment (day 0) will be carried out for 2 hours and ideally within 24 hours but not later than 48 hours after diagnosis of severe sepsis. The second PMX treatment has to be performed 24 to 48 hours after the end of the first PMX treatment, ideally after 24 hours. Hemoperfusion therapy will be performed in addition to conventional medical therapy in the ICU.
  Other Names: Toraymyxin
  Arms: 1
Other: Conventional medical therapy in the ICU — Including, but not limited to: antibiotic therapy, nutrition, administration of gamma-globulins, vasopressors, hemodynamic monitoring, organ support in the ICU including mechanical ventilation, corrective measures for metabolic abnormalities, renal replacement therapy when appropriate.

SUMMARY:
This clinical study designed as a prospective, open labelled, multi-centre, RCT will be carried out to evaluate if direct hemoperfusion with polymyxin B immobilized fiber column (PMX) is superior to conventional medical therapy for sepsis, for patients with sepsis arising from abdominal cavity infection, accompanied by the failure of one or more organs. 120 patients (60 treatment/60 control) will be considered in this study. Those patients fulfilling inclusion criteria and not having exclusion criteria will be randomly allocated to one of two study groups. One group will be treated with PMX (PMX group) and the other will receive a "standard therapy" for sepsis (control group). All patients will receive full intensive care management, including fluid resuscitation, vasopressors, antimicrobial chemotherapy, ventilatory support, and renal replacement therapy, if required. Each patient will be followed up for 28 days after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis due to intra-abdominal cavity infection after emergency surgery with at least 2 SIRS criteria and 1 organ dysfunction (as defined by SCCM)

Exclusion Criteria:

* Less than 18 years of age
* Females with a positive pregnancy test
* Treated with another investigational drug or device within the 30 days immediately preceding enrolment in this study
* Undergone organ transplantation during the past one year
* Documented history of sensitivity to Polymyxin-B, anticoagulant (heparin)
* Terminally ill, including metastases or hematological malignancy, with a life expectancy less than 30 days (as assessed by the attending physician) or have been classified as "Do Not Resuscitate"
* Diagnosed with HIV
* Previous history of end stage chronic organ failure(s)
* Uncontrolled hemorrhage within the last 24 h
* Diagnosed with granulocytopenia (leukocyte count of less than 500 cells/mm3) and/or thrombocytopenia (platelet count of less than 30,000 cells/mm3)
* More than 4 failed organs at entry
* An APACHE II score of more than 30 at entry to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure and use of vasopressors | 48-72 hrs

SECONDARY OUTCOMES:
PaO2/ FiO2 ratio | 48-72 hrs
Change in SOFA score | 48-72 hrs
ICU survival | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- St Bortolo Hospital, Vicenza, Italy

REFERENCES:
- [Background] Cruz DN, Perazella MA, Bellomo R, de Cal M, Polanco N, Corradi V, Lentini P, Nalesso F, Ueno T, Ranieri VM, Ronco C. Effectiveness of polymyxin B-immobilized fiber column in sepsis: a systematic review. Crit Care. 2007;11(2):R47. doi: 10.1186/cc5780. PMID 17448226
- [Derived] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784